CLINICAL TRIAL: NCT06386094
Title: Cirrhotic Cardiomyopathy and Cardiac Dysfunction in Patients with Metabolic Dysfunction Associated Steatotic Liver Disease
Brief Title: Cardiac Dysfunction in Patients with Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2023/SPL-902; IEC/2024/1523 dt 3.12.2024 (Other: Postgraduate Institute of Medical Education and Research)
Record Dates: First submitted 2023-09-19; First posted 2024-04-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: NAFLD; Cardiac Disease; Fatty Liver; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: MASLD; Cirrhotic Cardiomyopathy; Heart failure in Cirrhosis; Coronary Artery Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Heart Diseases; Fatty Liver; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MASLD: Non invasive tests like APRI, FIB-4, , FAST scan and VCTE in the form of Fibroscan will be done and recorded.
  Liver biopsy would be done as per the clinical indication. Diagnosis of NAFLD will be based on history, physical examination, laboratory investigations, upper gastrointestinal endoscopy, imaging studies (ultrasonography and Doppler of spleno portal venous axis, VCTE) and liver biopsy where available.
  Interventions: Diagnostic Test: Echocardiographic assessment

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment — M mode, cross sectional and pulsed wave Doppler Echocardiographic examinations will be performed using a with a 2.5 MHz wide angle phased array transducer. Patients will be laid in left lateral position and examined in standard parasternal long and short axis and apical views. Short axis recordings will be performed at the level of the papillary muscles. M mode tracings will be recorded at the level of the papillary muscles and the aortic valves, with 2 -D guidance. LV wall thickness and cavity diameters will be measured by M mode, through the largest diameter of the ventricle, if possible, both in diastole and systole. Using the cross-sectional images as a guide, the M mode tracing of the left ventricle will obtained to calculate measurements according to the recommendations of American Society of Echocardiography.

SUMMARY:
Cirrhotic cardiomyopathy is seen as a blunted contractile responsiveness to stress, and/or altered diastolic relaxation with electrophysiological abnormalities, in absence of known cardiac disease. Left ventricular diastolic dysfunction (LVDD) is associated with risk of hepatorenal syndrome (HRS) , septic shock. , heart failure in the perioperative period following liver transplantation, and after trans-jugular intrahepatic portosystemic shunt (TIPS) insertion . The echocardiographic E/e' ratio is a predictor of survival in LVDD, with multiple studies, including prospective data from our Centre. The inability of the heart to cope with stress or sepsis induced circulatory failure is a key concept of the increased mortality risk due to LVDD. In view of the metabolic syndrome and diabetes epidemic and an increasing number of patients being diagnosed with non-alcoholic fatty liver disease, there is increased risk of developing cardiac dysfunction due to multiple comorbidities including coronary artery disease, hypertensive heart disease, cirrhotic cardiomyopathy, which are contributors to overall cardiovascular risk of mortality.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) and heart failure (HF) are obesity-related conditions with high cardiovascular mortality. Many new studies have linked NAFLD to changes in myocardial energy metabolism, and to echocardiographic measurements of cardiac dysfunction especially heart failure with preserved ejection fraction. Cardiac dysfunction in NAFLD is related to the release of inflammatory cytokines among those with steatohepatitis (NASH). However composite models looking at coronary artery disease, systolic and diastolic heart failure and outcomes in patients with NAFLD are limited, and the few preliminary analyses of this relationship using histologically-defined NASH or lean NAFLD remain unclear.

In this project the investigators will screen patients with a diagnosis of 'non-alcoholic fatty liver disease' for presence of coronary artery disease, arrhythmias, cirrhotic cardiomyopathy and develop a model for cardiac dysfunction in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-65 years
* metabolic dysfunction associated steatotic liver disease as diagnosed either by histology or clinical, laboratory, non invasive tests, USG findings and vibration controlled transient elastography (VCTE).

Exclusion Criteria:

* Age >65 years
* Chronic renal disease
* Pregnancy and peripartum cardiomyopathy
* Hypertension
* Valvular heart disease
* Sick sinus syndrome/ Pacemaker
* Cardiac rhythm disorder
* Hypothyroidism
* Hyperthyroidism
* Portal vein thrombosis
* Transjugular intrahepatic porto systemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Anemia Hb < 8gm/dl in females, and < 9 gm/dl in males at the time of assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is all patients with a diagnosis of metabolic dysfunction associated steatotic liver disease seen in the outpatient and inpatient services of the Department of Hepatology, PGIMER Chandigarh.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of cardiac dysfunction in patients with non-alcoholic fatty liver disease/ metabolic dysfunction associated steatotic liver disease | At Enrolment
  Prevalence of CCM in the MASLD cohort

SECONDARY OUTCOMES:
Presence of myocardial abnormalities in CCM dysfunction | At Enrolment
  Use of cardiac MRI or CT
Presence of perfusion abnormalities in CCM dysfunction | At Enrolment
  Use of LV scintigraphy
All cause mortality in metabolic dysfunction associated steatotic liver disease | 12 months after enrolment
  All cause mortality will be recorded
Cardiac event related mortality in MASLD | 12 months after enrolment
  Cardiovascular events like incidence of arrhythmia, symptomatic heart failure related deaths will be recorded.
To determine the severity of cardiac dysfunction in patients with metabolic dysfunction associated steatotic liver disease | At Enrolment
  Prevalence of CCM in the MASLD cohort, and grade of LV diastolic and systolic dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Madhumita Premkumar, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365